CLINICAL TRIAL: NCT04914767
Title: The Effectiveness of Nigella Sativa in the Treatment of SARS COV2 (COVID-19)
Brief Title: Nigella 5 in the Treatment of SARS COV2 (COVID-19)
Acronym: Nigelle5
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hôpital Universitaire Sahloul (Other)
Responsible Party: Principal Investigator, Riadh Boukef, PROFESSOR, Hôpital Universitaire Sahloul
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NigCOV1&2
Record Dates: First submitted 2021-05-28; First posted 2021-06-07 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19 | interventions — Nigella sativa oil

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nigella (Experimental): The patient will receive a study treatment containing 100 capsules:
  * One capsule every two hours for the first three days.
  * From the fourth day, the patient will take one capsule, three times a day for 12 days.
  Interventions: Drug: Nigella
- Placebo Group (Placebo Comparator): The patient will also receive a study treatment containing 100 capsules:
  * One capsule every two hours for the first three days.
  * From the fourth day, the patient will take one capsule, three times a day for 12 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nigella — The patient will receive a study treatment containing 100 capsules:
  * One capsule every two hours for the first three days.
  * From the fourth day, the patient will take one capsule, three times a day for 12 days.
  Arms: Nigella
Drug: Placebo — The patient will receive a study treatment containing 100 capsules:
  * One capsule every two hours for the first three days.
  * From the fourth day, the patient will take one capsule, three times a day for 12 days.
  Arms: Placebo Group

SUMMARY:
The world is currently facing a crisis because of this potentially fatal situation of the COVID-19 epidemic without proven efficacy for any drug treatment, while the vaccination is not yet.

This epidemic is caused by a new betacorona virus, now called SARS-CoV-2. The most common symptoms reported are fever, cough or chest tightness, and dyspnea. Most cases have a mild course

DETAILED DESCRIPTION:
In the absence of proven antiviral therapy or specific vaccination against COVID-19, Nigella seed oil is suggested as a potential supplement due to its known immunostimulatory and antiviral activities in previous published studies.

Nigella (known as black seed) in the Latin language or "Habatulbarakah" in the Arabic language, is a food supplement and a medicinal plant well known in Arab and Islamic culture. It is used as a food spice and it has a lot of medical claims that come from different historical backgrounds. Nigella seeds contain several active compounds that have been isolated, identified and reported, the most important being thymoquinone.

In the literature, black seed has shown several pharmacological activities, including anti-inflammatory, antiviral and immunostimulatory activities.

ELIGIBILITY:
Inclusion Criteria: patients included in the two studies NIGCOV1 and NIGCOV2 must be:

* Men and women at least 40 years old, able and willing to give informed consent;
* Ambulatory (NIGCOV1) or hospitalized (NIGCOV2) environment;
* Patient with dyspnea or with a positive gait test (NIGCOV2);
* The patient must have at least one of the following high risk criteria: 70 years or older, obesity (BMI ≥ 30 kg / m2), diabetes mellitus, uncontrolled hypertension (systolic blood pressure ≥ 150 mm Hg), respiratory disease known (including asthma or chronic obstructive pulmonary disease), known heart failure, known coronary artery disease, fever ≥ 38.4 ° C within the last 48 hours, dyspnea at the time of presentation (only patients included on NIGCOV2), bicytopenia, pancytopenia or a combination of a number high neutrophils and low lymphocytes count (only patients included on NIGCOV2);
* The patient is not of childbearing age, defined as postmenopausal for at least 1 year or surgically sterile, or is of childbearing age and uses at least one method of contraception and preferably two complementary forms of contraception comprising a method of barrier throughout the study and for 30 days after the end of the study;
* The patient must be able and willing to comply with the requirements of this study protocol.

Exclusion Criteria:

* Patient currently in shock or exhibiting hemodynamic instability;
* Patient with inflammatory bowel disease (Crohn's disease or ulcerative colitis), chronic diarrhea or malabsorption;
* Pregnant or breastfeeding patient
* Patient with a history of allergic reaction or significant sensitivity to Nigella;
* The patient is considered by the investigator, for whatever reason, to be an unsuitable candidate for the study.

Given the non-homogeneity of the patients, the study population will be divided into two groups:

* group of outpatients: Ambulatory patients = NIGCOV1 study
* and inpatient group: Hospitalised patients = NIGCOV2 study Statistical analysis will be carried out for each group separately

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of Death or readmission or requiring oxygen supplementation | one months
  The composite of death or need for hospitalization or requiring oxygen supplementation due to COVID-19 infection within the first 30 days of randomization

SECONDARY OUTCOMES:
Death Rate | one month
  The occurrence of death within 30 days of randomization
Rate of Requiring oxygen supplementation | one month
  Number of participants requiring oxygen supplementation
Rate of Hospiatalization | one month
  Number of participants requiring hospitalization due to COVID19 infection

CONTACTS AND LOCATIONS:
Overall Officials: Riadh Boukef, professor, Principal Investigator — CHU Sahloul, Sousse, Tunisia
Locations (2):
- Tunisia (2):
  - HU Sahloul, sousse, Tunisia, Sousse, Itinéraire Ceinture Cité Sahloul
  - Riadh Boukef, Sahloul, Sousse Governorate

IPD SHARING:
Plan to Share IPD: No
in the article publication